CLINICAL TRIAL: NCT06621524
Title: Coronary Angioplasty With Sirolimus Drug-coated Stent System to Treat Patients With Symptomatic Ischemic Coronary Heart Disease: a PMCF Study.
Brief Title: EucaLimus Post-Market Registry
Status: Active, not recruiting | Type: Observational
Sponsor: OrbusNeich (Industry)
Collaborators: Eucatech AG (Industry); Centre Européen de Recherche Cardiovasculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: DVAL-PLAN-0062
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Coronary Arterioscleroses
Keywords: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases; Drug-Coated Stent; Ischemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device: EucaLimus coronary stent system: The EucaLimus coronary stent system is a drug-coated coronary stent system, indicated for use in patients with symptomatic ischaemic coronary heart disease due to de novo lesions or restenosed lesions of the coronary arteries.
  Interventions: Device: EucaLimus coronary stent system

INTERVENTIONS:
Device: EucaLimus coronary stent system — The EucaLimus coronary stent system is a drug-coated coronary stent system, indicated for use in patients with symptomatic ischaemic coronary heart disease due to de novo lesions or restenosed lesions of the coronary arteries.

SUMMARY:
To collect post marketing surveillance data on consecutive patients with coronary heart disease intended to be or treated by the Eucalimus sirolimus eluting PTCA stent when used according to the Instructions for Use. Data will be collected in order to assess the long term safety and performance of the Eucalimus PTCA stent in routine clinical practice.

DETAILED DESCRIPTION:
The multicenter, prospective registry population consists of consecutive patients with coronary heart disease who undergo percutaneous coronary intervention (PCI) and are intended to be or treated by the Eucalimus sirolimus eluting PTCA stent (according to the Instructions for Use) as part of routine clinical care. Approximately 251 patients from 5-10 centers in Europe and Asia will be entered into the registry. Patients entered into the registry are followed for three years. The registry is considered finished when all patients have completed the 36-month follow-up.

A follow-up is scheduled at the following timepoints: immediately post-procedure, 30 days, 6 months, 12 months, 24 months, and 36 months. Follow-up is obtained by telephone contact with the patient or at a planned hospital visit.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients intended to be, or treated by EucaLimus as per physicians' decision and according to Instructions for Use (IFU) in the setting of routine clinical care are entered into the registry.

Exclusion Criteria:

* Patients are excluded from registration if ANY of the following conditions apply:

  * High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
  * Currently participating in another investigational drug or device study in which a routine angiographic follow-up is planned
  * A life expectancy of <1year
  * Explicit refusal of participation in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic ischaemic coronary heart disease due to de novo lesions or restenosis lesions of the coronary arteries, or patients with acute or suspected occlusions who responded unsuccessfully to an interventional therapy following balloon dilatation.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Adjudicated, device-oriented, Target Lesion Failure (TLF) | 12 months post procedure
  Adjudicated, device-oriented, Target Lesion Failure (TLF) where TLF is defined (Academic Research Consortium- ARC) as a composite of cardiac death (CD), non-fatal myocardial infarction (MI) not clearly attributable to a non-target vessel (TV-MI) or clinically driven target lesion revascularization (cd-TLR).

SECONDARY OUTCOMES:
Adjudicated Target Lesion Failure (TLF) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Each of the components of TLF (Cardiac Death (CD), non-fatal myocardial infarction not clearly attributable to a non-target vessel (TV-MI), clinically driven target lesion revascularization (cd-TLR)) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated Target Vessel Failure (TVF) (ARC definition) as a composite of Cardiovascular Death (CVD), TV-MI and clinically driven target vessel revascularization (cd-TVR) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Each of the components of TVF (Cardiovascular Death (CVD), TV-MI and clinically driven target vessel revascularization (cd-TVR)) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated stent thrombosis per ARC-2 definition | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated bleeding Type 3-5 per the Bleeding Academic Research Consortium (BARC) definition | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated stroke | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Device success | Index Procedure
  Device success: Percentage of patients with a successful delivery and deployment of the EucaLimus stent at the target lesion and final diameter stenosis after stenting ≤20% by visual assessment in the presence of grade 3 TIMI (Thrombolysis in Myocardial Infarction) flow, by visual estimation EucaLimus stent at the target lesion and a final diameter stenosis after stenting ≤20% by visual assessment in the presence of grade 3 TIMI flow, by visual estimation
Procedure Success | Index Procedure
  Procedure Success: Device success and no peri-procedural death, MI or TVR.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Gomez-Lara, MD, PhD, Principal Investigator — Bellvitge University Hospital
Locations (10):
- Czechia (2):
  - Krajska nemocnice Liberec, Liberec
  - Motol University Hospital, Prague
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Spain (7):
  - Bellvitge University Hospital, L'Hospitalet de Llobregat, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo
  - Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No